CLINICAL TRIAL: NCT04606290
Title: Automated Oxygen Titration to Patients with COPD and Domiciliary Long-term Oxygen Treatment
Brief Title: Automated Oxygen Titration with O2matic Home Oxygen Therapy (O2matic HOT) Phase 1
Acronym: O2matic-HOT1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual); Naestved Hospital (Other)
Responsible Party: Principal Investigator, Ejvind Frausing Hansen, Chief Physician, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: O2matic-HOT1
Record Dates: First submitted 2020-10-24; First posted 2020-10-28 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: COPD; Chronic Hypoxemic Respiratory Failure
Keywords: O2matic; Closed-loop; Pulse oximetry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Manual (Active Comparator): Fixed dose oxygen
  Interventions: Device: Oxygen concentrator
- O2matic (Experimental): Automated oxygen titration
  Interventions: Device: O2matic HOT

INTERVENTIONS:
Device: O2matic HOT — Automated oxygen titration with O2matic HOT
  Arms: O2matic
Device: Oxygen concentrator — Fixed dose oxygen flow from concentrator
  Arms: Manual

SUMMARY:
O2matic HOT is a further development of O2matic and is intended for home oxygen use with patients in need of long-term oxygen treatment (LTOT). O2matic HOT is a closed-loop system which on basis of signals from pulse oximetry titrates the oxygen flow to the patient. In this crossover trial patients are admitted for 24 hours twice. Once with usual fixed dose oxygen and once with oxygen titration by O2matic HOT.

DETAILED DESCRIPTION:
The purpose of this study is to examine if automated oxygen control based on pulse oximetry to patients with domiciliary long-term oxygen treatment (LTOT) is better than manually controlled oxygen treatment in keeping SpO2 within intended target interval. In manually controlled oxygen treatment flow is usually kept constant for months between visits from specialist nurse, whereas in automated control the patient can titrate oxygen flow several times a day based on pulse oximetry in a closed-loop system.

ELIGIBILITY:
Inclusion Criteria:

* Verified COPD with FEV1/FVC < 0.70
* Need of LTOT (PaO2 <= 7.3 kPa or SpO2 < 88 % on ambient air)
* Cognitively able to participate
* Willing to provide informed consent

Exclusion Criteria:

* Moderate or severe exacerbation in COPD within 4 weeks from study start
* Major comorbidities (cancer, uncontrolled chronic disease)
* Asthma or other disease with need of higher SpO2
* Pregnancy
* Fall in pH below 7.35 or increase in PaCO2 > 1 kPa on 5 liters of oxygen
* Active smoking
* LTOT use less than 1 hours/day

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of time in intended SpO2-interval | 24 hours
  Percentage of time with SpO2 in intended interval

SECONDARY OUTCOMES:
Percentage of time with SpO2 below 85 % | 24 hours
  Percentage of time with SpO2 below 85 %
Percentage of time with SpO2 below target but not below 85 % | 24 hours
  Percentage of time with SpO2 below target but not below 85 %
Percentage of time with SpO2 above target | 24 hours
  Percentage of time with SpO2 above target
Change in PaCO2 from baseline | 8 hours
  Change in PaCO2 from baseline to 8 hours
Change in PaCO2 from baseline | 24 hours
  Change in PaCO2 from baseline to 24 hours
Accumulated oxygen usage | 24 hours
  Accumulated oxygen usage in 24 hours
Adverse and serious adverse events | 24 hours
  Adverse and serious adverse events, such as respiratory acidosis

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ringbaek, PhD, Study Chair — Hvidovre University Hospital
Locations (2):
- Denmark (2):
  - Hvidovre University Hospital, Hvidovre
  - Næstved University Hospital, Næstved

IPD SHARING:
Plan to Share IPD: No